CLINICAL TRIAL: NCT01120808
Title: Prevention Trial Assessing Paper-Tape in Endurance Distances (PreTAPED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of California, Davis (Other)
Responsible Party: Principal Investigator, Grant S Lipman, PI, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SU-04282010-5782
Record Dates: First submitted 2010-05-07; First posted 2010-05-11 (Estimated); Results first posted 2017-03-24 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-11

CONDITIONS: Blister
MeSH Terms: conditions — Blister

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All Participants (Experimental): Participants were registered competitors in RacingThePlanet 6 stage 7 day 155mile (250km) ultramarathon.
  Interventions: Procedure: Paper tape

INTERVENTIONS:
Procedure: Paper tape — Paper tape assigned to each participant's randomly selected foot.

SUMMARY:
Blisters are a very common complaint in both the general population and also the athlete. This study's aim is to determine whether applying paper tape (an inexpensive and common component of most foot care kits) to the foot of endurance runners prevents the frequency and severity of friction blisters.

DETAILED DESCRIPTION:
Participants will be approximately 100 ultra-endurance athletes competing in Racing the Planet's 250 mile/7 day 4 Desert ultra-endurance races. A convenience sample will be used, with full consent signed before inclusion into the study, with participants being informed that study inclusion is entirely optional and will not affect medical care. A foot will berandomly selected for each participant, a coin will be flipped to determine which foot is to be taped, heads - right foot, and tails, left foot. The non-taped foot will be used as a control. No preventive treatment will be applied to the control foot. The runner's normal sock/shoe system will be used to reflect natural wilderness conditions. Runners will be excluded if any blisters, broken blisters, or hot spots are present on either foot at the time of initial taping as determined by visual foot inspection by a study administrator. The participant will also be excluded if they have a pre-existing blistering condition or known sensitivity to paper tape. Participants will have demographic data collected prior to the race, including age, gender, country of origin, number of marathons run prior, pack weight, and sock type. The study endpoint occurs when a hot spot or blister develops on either the treated or untreated foot. Runners will be instructed to treat suspected blisters or hot spots as they normally would, and to inform the study administrators the same day for visual inspection and final questionnaire to determine if they develop blisters or hot spots, whether they applied or re-applied tape themselves, removed tape, and the reasons for these actions. Participants will be allowed to have their experimental taped foot re-taped by a physician at any point in the race as deemed necessary by the runner. Before applying tape, a visual inspection will determine that feet were clean of dirt and no hot spots or blisters / broken blisters were present. Tape will be applied by trained study physicians. One inch micropore paper tape from 3M will be applied to each toe in the following manner. A piece of tape will be placed on each toe longitudinally from the base of the phalanx dorsally to the base of the phalanx on the plantar side. The tape will be smoothed against the skin. Any tape extending beyond the tip of the phalanx will be adhered together. A second piece of one inch paper tape will be applied circumferentially around each toe, with the ends of the tape located on the dorsum of the toe. In this manner, all five toes on the experimental foot will be taped. Any "dog ears" (tape extending beyond the phalanges) will be then trimmed with a scissors. One 2 inch piece of micropore paper tape will be applied horizontally to the posterior heel over the Achilles tendon, extending from the posterior medial malleolus to the posterior lateral malleolus. One 2 inch piece of micropore tape will be applied perpendicular to the head of the 5th metatarsal, another perpendicular to the 1st metatarsal covering medial as well as plantar aspect.

ELIGIBILITY:
Inclusion Criteria:

* All runners who are enrolled in an RTP 4 deserts event,
* All runners who are 18-75 years old, and
* All runners who speak English. The study will be enrolling only those who speak English, so they can fully understand and have knowledgeable consent to the study enrollment protocols.

Exclusion Criteria:

* Any blisters, broken blisters, or hot spots present on either foot at the time of initial taping as determined by visual foot inspection by a enrolling study physician.
* The runner has a pre-existing blistering condition.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2010-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grant S Lipman, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - University of California Davis, Davis, California
  - Stanford University School of Medicine, Stanford, California

REFERENCES:
- [Result] Lipman GS, Ellis MA, Lewis EJ, Waite BL, Lissoway J, Chan GK, Krabak BJ. A prospective randomized blister prevention trial assessing paper tape in endurance distances (Pre-TAPED). Wilderness Environ Med. 2014 Dec;25(4):457-61. doi: 10.1016/j.wem.2014.06.013. Epub 2014 Oct 31. PMID 25443754

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants
Started | 136
Completed | 90
Not Completed | 46

BASELINE CHARACTERISTICS:
Population: Per protocol, participants completing the primary outcome measure were analyzable for baseline characteristics.
Arm/Group | All Participants
Number analyzed (Participants) | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 58

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants With Blisters
Time Frame: 1 week
Population: Participants with available data were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 90
Participants
  Blisters on both feet | 8
  Blister on taped foot | 47
  Blister on untaped foot | 35

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/90
Other Adverse Events (participants affected / at risk) | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No